CLINICAL TRIAL: NCT01856569
Title: Assial - Anti Tnf Treatment In Ankylosing Spondylitis: An Observational Cohort Study In Italy
Acronym: ASSIAL
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801362; B1801362
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — in real life of drug,dosage,frequency and duration
  Other Names: adherence of therapy,switching,combo therapy

SUMMARY:
Observe in real life adherence therapy and time to switch in ankylosing spondylitis patients with predominant assial involvement with 4 anti-TNF.

DETAILED DESCRIPTION:
retrospective and prospective 150

ELIGIBILITY:
Inclusion Criteria:

retrospective:12 months at least first anti-TNF therapy prospective: at maximum 6 months observation AS patients with axial involvement

Exclusion Criteria:

patients in other AS studies involved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ankylosing spondylitis
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Italy (18):
  - Unita Operativa Semplice di Reumatologia, Catania, CT
  - Arcispedale Sant'Anna, Ferrara, Italy
  - U.O.S. Reumatologia - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola-Malpighi, Bologna
  - Piazzale Spedali Civili, Brescia
  - Policlinico Di Cagliari, Dipartimento Di Scienze Mediche, Cagliari
  - Via Torregalli, 3, Florence
  - Ospedale Ortopedico G. Pini, Milan
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Policlinico Universitario, II Universita, Napoli
  - Policlinico Universitario, Padua
  - Divisione di Reumatologia, Palermo
  - Policlinico Universitario P. Giaconne, Palermo
  - Azienda USL 4 di Prato, Prato
  - Università Campus Bio-Medico di Roma- Policlinico Universitario Campus Bio-medico di Roma, Roma
  - Policlinico Umberto I, Roma
  - Ospedale Mauriziano Umberto I, Torino
  - Policlinico Universitario, Udine
  - Ospedale Borgo Trento - Clinica Reumatologica, Verona

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801362&StudyName=Assial%20-%20Anti%20Tnf%20Treatment%20in%20Ankylosing%20Spondylitis%3A%20an%20Observational%20%20Cohort%20Study%20in%20Italy%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-Tumor Necrosis Factor (Anti-TNF): Participants with ankylosing spondylitis (AS), who had started the anti-TNF-alpha treatment (as per physician's discretion based on summary of product characteristics) for at least 12 months prior to enrollment, were followed up to 18 months.
Period: Overall Study
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Started | 152
Full Analysis Set | 144
Completed | 139
Not Completed | 13
Not completed — Other | 1
Not completed — Changed Site/Structure | 1
Not completed — Lost to Follow-up | 3
Not completed — Did not met inclusion criteria | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who met the inclusion criteria.
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.85 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Unchanged First Line Anti-TNF Treatment Up to Month 18
Description: First line anti-TNF treatment included adalimumab, etanercept, golimumab and infliximab. In this outcome, percentage of participants who were taking any one of the first line anti-TNF treatment at baseline and maintained the same up to Month 18 without any change in prescription, were reported.
Time Frame: Baseline up to Month 18
Population: FAS included all participants who met the inclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 144
percentage of participants | 85.42

2. Primary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Month 18
Description: BASDAI was a validated self-assessment tool used to determine disease activity in participants with AS. Utilizing a numerical rating scale (NRS) of 0-10 (0 = no problem to 10 = worst problem) participants answered 6 questions measuring symptoms of AS (spinal pain, fatigue, joint pain or swelling, areas of localized tenderness, morning stiffness duration and severity). The BASDAI total score was calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score was then divided by 5. BASDAI=Q1+Q2+Q3+Q4+[Q5+Q6/2]/5. The total BASDAI score ranges from 0=none to 10=severe, where lower score indicated less disease activity.
Time Frame: Baseline, Month 18
Population: FAS included all participants who met the inclusion criteria. Here, number of participants analyzed (N) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 113
units on a scale | 3.84 (2.41)

3. Primary Outcome: Percentage of Participants With Unchanged First Line Anti-TNF Treatment In State of Low Disease Activity
Description: Low disease activity was defined as a BASDAI score of less than or equal to (<=) 2. BASDAI was a validated self-assessment tool used to determine disease activity in participants with AS. The total BASDAI score ranges from 0=none to 10=severe, where lower score indicated less disease activity. In this outcome, percentage of participants with unchanged first line anti-TNF drug (nor dose neither frequency, but drug only) in the state of low disease activity, during the specified time points were reported.
Time Frame: Month 12, 18
Population: FAS included all participants who met the inclusion criteria. Here, "n" signifies number of participants evaluable for each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 144
percentage of participants
  Month 12 (n=65) | 60.19
  Month 18 (n=73) | 61.86

4. Secondary Outcome: Ankylosing Spondylitis Quality of Life (ASQoL) Total Score at Month 18
Description: ASQoL was a disease-specific questionnaire that assessed the impact of AS on participant's quality of life (QoL). It consisted of 18 questions to be completed by the participant. Each question was answered by the participant as a 'Yes' (scored as 1) or 'No' (scored as 0). Scores of each individual question was summed to give a total score that ranges from 0 (good QoL) to 18 (poor QoL), where lower scores indicated good quality of life. Data for this outcome was planned to be reported separately for switchers (participants who switched to a second anti-TNF drug during observation period) and non-switchers (participants who did not switched to a second anti-TNF drug during observation period).
Time Frame: Month 18
Population: FAS included all participants who met the inclusion criteria. Here, "n" signifies number of participants evaluable each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 144
units on a scale
  Switchers (n= 21) | 5.4 (4.7)
  Non-switchers (n= 123) | 3.0 (4.2)

5. Secondary Outcome: C Reactive Protein Level at Baseline
Description: C reactive protein was measured from blood samples as a marker for inflammation. Higher levels were indicative of more inflammation.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram per liter
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 141
milligram per liter | 5.91 (10.53)

6. Secondary Outcome: Erythrocyte Sedimentation Rate at Baseline
Description: Erythrocyte sedimentation rate was a laboratory test that provided a non-specific measure of inflammation. The test assessed the rate at which red blood cells fell in a test tube and was measured in millimeter per hour (mm/h).
Time Frame: Baseline
Population: FAS included all participants who met the inclusion criteria.
Measure: Mean (Standard Deviation); unit: millimeter per hour
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Number analyzed (Participants) | 144
millimeter per hour | 25.91 (19.64)

ADVERSE EVENTS:
Arm/Group | Anti-Tumor Necrosis Factor (Anti-TNF)
Serious Adverse Events (participants affected / at risk) | 0/144
Other Adverse Events (participants affected / at risk) | 28/144
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-Tumor Necrosis Factor (Anti-TNF) (N=144)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Gastroenteritis viral (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Hypersensitivity (Immune system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Migraine (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Injection site erythema (General disorders) | 3
Chest pain (General disorders) | 1
Infusion site urticaria (General disorders) | 1
Conjunctivitis viral (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Data for change from baseline in ASQoL score was not collected as per change in planned analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.